CLINICAL TRIAL: NCT01728688
Title: Safety and Efficacy of Human Autologous Peripheral Blood Stem Cells for Treatment of HBV-related Liver Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Eastern Hepatobiliary Surgery Hospital (Other); Chinese Academy of Medical Sciences (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Han Ying, professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120912-2
Record Dates: First submitted 2012-10-31; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Liver Cirrhosis; End Stage Liver Disease
Keywords: liver cirrhosis; stem cell; peripheral blood; autologous; HBV; end stage liver disease
MeSH Terms: conditions — Liver Cirrhosis; End Stage Liver Disease | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Active Comparator): conventional treatment & antiviral treatment
  Interventions: Other: conventional treatment
- conventional & PBSC transplantation (Experimental): After three days G-CSF mobilization, Patients randomized to the intervention arm will receive autologous PBSCs transplantation at day1, and receive conventional treatment and antiviral treatment through the one year study visit and followed until one years study visit.
  Interventions: Other: PBSC transplantation

INTERVENTIONS:
Other: PBSC transplantation — PBSCs were mobilized with recombinant human G-CSF at 5-10ug/kg/d for three days. then PBSCs were collected by means of apheresis. The collected PBSCs were infused into participant via hepatic artery
  Arms: conventional & PBSC transplantation
Other: conventional treatment — Participants will receive conventional treatment and antiviral treatment.
  Arms: Conventional

SUMMARY:
HBV related Liver disease is a common medical problem in China. An estimated 7.18% of the Chinese (about 93 million) is infected with hepatitis B, and most of the HBV- related hepatitis can developed into liver cirrhosis.

Liver transplantation is the only available life saving treatment for patients with end stage liver disease. However, lack of donors, surgical complications, rejection, and high cost are serious problems.

In preclinical studies the investigators have demonstrated that G-CSF mobilized PBSC from patients with HBV related liver cirrhosis could differentiate into functional hepatocyte and autologous PBSC transplantation can significantly improve liver synthetic function. But further studied was needed to confirm the safety and efficacy of PBSC transplantation. In this study, a prospective, randomized, parallel clinical study was designed. The patients with HBV-related liver cirrhosis will undergo administration of human autologous PBSCs via hepatic artery to evaluate the safety and efficacy of human autologous PBSCs treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. HBV-related liver cirrhosis
3. Child-Pugh score 9-15
4. Written consent

Exclusion Criteria:

1. Hepatocellular carcinoma or other malignancies
2. Severe problems in other vital organs(e.g.the heart,renal or lungs)
3. Pregnant or lactating women
4. Severe bacteria infection
5. Anticipated with difficulty of follow-up observation
6. Other candidates who are judged to be not applicable to this study by doctors -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
one-year survival rate | one year after treatment

SECONDARY OUTCOMES:
MELD score | 1week, 4weeks,3months, 6months, 9months and 1year after treatment
Child Pugh Score | 1week, 4weeks,3months, 6months, 9months and 1year after treatment
alpha fetoprotein | 1week, 4weeks,3months, 6months, 9months and 1year after treatment
renal function | 1week, 4weeks,3months, 6months, 9months and 1year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daiming Fan, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China